CLINICAL TRIAL: NCT05507021
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Lactobacillus Plantarum DSM 33464 (SmartGuard <TM>/MegametalliQ <TM>) to Reduce Blood Lead Levels in Young Women of Child-bearing Age (18 to 40 Years Old)
Brief Title: Effect of Lactobacillus Plantarum DSM 33464 on Blood Lead Levels in Young Women of Child-bearing Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: Universidad Iberoamericana A.C., Mexico (Other); Linus Biotechnology Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NZ-2021-03
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Elevated Blood Lead Levels
Keywords: Blood lead level; Lactobacillus Plantarum DSM 33464

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus plantarum DSM 33464, MegaMetalliQ (Experimental): Subjects will take 1 sachet of Lactobacillus plantarum DSM 33464 (2 g) per day for 8 weeks
  Interventions: Dietary Supplement: Lactobacillus plantarum DSM 33464, MegaMetalliQ
- placebo group (Placebo Comparator): Subjects will take 1 sachet of Placebo (2 g) per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum DSM 33464, MegaMetalliQ — Pour Lactobacillus Plantarum DSM 33464 sachet into moderate amount of water, slightly stir, fully dissolve, drink 0.5 hour before having meal, one at a time.
  Arms: Lactobacillus plantarum DSM 33464, MegaMetalliQ
Dietary Supplement: Placebo — Pour placebo sachet into moderate amount of water, slightly stir, fully dissolve, drink 0.5 hour before having meal, one at a time.
  Arms: placebo group

SUMMARY:
We hypothesize that Lactobacillus Plantarum DSM 33464 reduce lead levels. Approximately 200 women 18 to 40 will be screened for blood lead levels. From that pool of subjects, 40 healthy women aged 18 to 40 years will participate in this randomized, placebo controlled pilot clinical trial. Each participant will receive 1 sachet of Lactobacillus Plantarum DSM 33464 (2g) per day for 8 weeks. The participants will be evaluated for several health measures, e.g. Blood, urine and hair will be collected and analyzed for lead (Pb) as the primary target compound and other chemicals as secondary target compounds. Adverse events will be recorded throughout the trial. Stool samples will also be collected at the beginning and end of the study to undertake a microbiome analysis.

DETAILED DESCRIPTION:
Introduction: Lead (Pb) is a heavy metal, toxic to humans. Exposure to Pb has been associated with a wide range of adverse health effects and is one of the major environmental health problems in terms of the number of people exposed and the cost of the public health implications involved. However, a major limitation in the treatment of chronic Pb exposure is that there is no successful treatment to decrease absorption and increase excretion via the gastrointestinal tract, particularly when exposure occurs at medium and low levels where most of the population is concentrated.

Objective: To explore the efficacy of Lactobacillus plantarum DSM 33464 (SmartGuardTM/MegametalliQTM) in reducing blood lead (PbS) levels in women over an 8-week period.

Methods: Double-blind, randomized, placebo-controlled clinical trial. The study consists of two stages: screening and supplementation. In the first stage of the study, a participant selection process will be carried out for which 200 women between 18 and 40 years of age, residents of Colonia Santa Fe, Mexico City, will be invited to undergo screening procedures to identify those who meet the inclusion criteria of the study. From this group, 40 women will be selected to continue participating in the second stage of the clinical trial. Through randomization, the participants will be assigned to the control group (placebo) or treatment (SmartGuardTM/MegametalliQTM). The supplementation will last 8 weeks (2 months), each participant will be given a kit including a box with 40 sachets, the participant will receive one box at visit 1 and a second box at visit 2 (1 sachet per day, each sachet containing 2 g. of SmartGuardTM/MegametalliQTM or placebo). A total of 80 sachets will be given so that the participant will have extra sachets in case she does not attend the second visit at exactly 4 weeks, or if she misplaces them for any reason; however, it will be emphasized that only 1 sachet per day should be taken and the leftovers should be returned to the researcher in charge for their correct disposal and elimination. During the intervention period, 4 visits are planned (V1, V2, V3 and V4) in which blood, urine and hair samples will be collected and analyzed and used to quantify the levels of Pb (main objective) and other chemical substances (secondary objective). At visits V1 and V3, stool samples will be collected for microbiome analysis. Participants will then be monitored for a further 4 weeks to assess medium-term effectiveness, as well as to identify any subsequent complications, such as micronutrient depletion.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years old.
* Women with capillary blood Pb levels between 3.3 µg/dL (Lead Care detection limit) and 25 µg/dL.
* Residents of Santa Fe, Mexico City.
* Women of childbearing age, using the same contraceptive method (any) since at least 3 cycles before the start of the study and who agree to maintain it for the entire duration of the study.
* Women who give their informed consent in writing.

Exclusion Criteria:

* Women with a diagnosed history of diseases of the nervous system, genetic diseases, endocrine diseases, lung diseases, serious or uncontrolled cardiovascular diseases, clinically significant kidney or liver diseases, diseases of the blood system, any other clinically significant disease, and others that the investigators consider would increase the risk of disease of the subject.
* Pregnant or lactating women, who intend to become pregnant or who declare that they have intended to become pregnant within the previous 3 months.
* Consumption of nutritional supplements 4-6 weeks before screening.
* Consumption of probiotic or antibiotic products in the last two weeks.
* Women who have received chelation therapy for Pb poisoning.
* Known or suspected allergy or sensitivity to study products or any component tested in the trial.
* Participation in another clinical trial or food study 4 weeks before and during the trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — • Women between 18 and 40 years old.
Enrollment: 47 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Blood Lead levels | 8 weeks
  Evaluate the effect of L. plantarum DSM 33464 to reduce the levels of blood lead in women during a period of 8 weeks in comparison with the ingestion of placebo.

SECONDARY OUTCOMES:
Blood lead levels | 4 weeks
  Evaluate the change in blood lead levels in response to ingestion of DSM 33464 (MegaMetalliQ<TM>)in participating women during the supplementation period compared to women in the placebo group.
Hair lead levels | 4 and 8 weeks
  Evaluate the change in hair lead levels in response to ingestion of DSM 33464 in participating women during the supplementation period compared to women in the placebo group.
Profile of heavy metal elements in the hair | 4 and 8 weeks
  The elements to be measured are Mg, P, S, Ca, Cr, Cu, Zn, Sr, Sn, I, Ba, Li, Al, Mn, Fe, Co, Ni, As, Cd, Hg, Bi, with the same unit g/dL
Composition of fecal microbiota | 8 weeks
  The composition of fecal microbiota will be measured in response to ingestion of DSM 33464 compared to ingestion of placebo.
Profile of heavy metal elements in the blood | 4 and 8 weeks
  The elements to be measured are Ca, Fe, Zn, Mg, Co, with the same unit g/dL
Profile of heavy metal elements in the urine | 4 and 8 weeks
  The elements to be measured are summarized in the protocol, examples are Bisphenol A and Butyl Paraben with the same measurement unit
Number of participants with intervention-related adverse events as assessed by CTCAE v4.0 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra de Jesús Cantoral Preciado, Ph.D, Principal Investigator — Universidad Iberoamericana A.C.
Locations (1):
- Universidad Iberoamericana A.C., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No